CLINICAL TRIAL: NCT02638675
Title: Examining Financial Health Incentives to Promote Physical Activity Among Inactive Hospital Employees: A Web-based Randomized Control Trial
Brief Title: Financial Health Incentives to Promote Physical Activity Among Hospital Employees: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Green Shield Canada Inc. (Industry); Cookson James Loyalty Inc. (Industry); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Guy Faulkner, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C4L-01
Record Dates: First submitted 2015-12-16; First posted 2015-12-23 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Physically Inactive Hospital Employees
Keywords: financial health incentives; physical activity; behavioral economics; randomized control trial; workplace health
MeSH Terms: conditions — Motor Activity | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wellness program, accelerometer, incentives (Experimental): During the intervention period (weeks 1 to 12), intervention participants will be eligible to earn daily reward points contingent on step count goal achievement. Intervention participants will earn 100 reward points (i.e. $1) for each day that specific step count goals are reached. During weeks 13 to 24, participants will no longer receive daily reward points for completing specific step count goals.
  Interventions: Behavioral: Wellness program; Device: Accelerometer; Behavioral: Incentive
- Wellness program and accelerometer (Active Comparator): During the 24 week trial, control participants will receive no additional incentives when step count goals are reached.
  Interventions: Behavioral: Wellness program; Device: Accelerometer

INTERVENTIONS:
Behavioral: Wellness program — All participants have access to Change4Life, a web-based health education and behaviour change program. Individuals are rewarded with very modest incentives (uncertain chance; less than 1 in 100 chance of earning) when they complete learning modules or health tasks.
Device: Accelerometer — All participants will be asked to wear the StepsCount Piezo accelerometer, which tracks steps and bout minutes of MVPA per day, synchronize the device to the Change4Life program, and reach daily step count goals for 24 weeks.
Behavioral: Incentive — During the first 12 weeks, participants will be eligible to earn $1 in vouchers (e.g., grocery, cinema) when daily goals are reached. The total amount available over the 3-month intervention period will be $90 (9,000 points). During weeks 13 to 24, participants will not receive daily reward points for completing step count goals.
  Arms: Wellness program, accelerometer, incentives

SUMMARY:
The objective of this randomized control trial is to examine whether incentives-for-steps (i.e. $1 per day step count goals are reached) increase daily step counts among physically inactive hospital employees.

DETAILED DESCRIPTION:
A 24-week, parallel arm, randomized control trial will be employed to examine the impact of incentives on physical activity among physically inactive Hamilton Health Science Corporation employees. Participants will be randomly allocated (1:1) into control (i.e. wellness program and accelerometer) or intervention groups (i.e. wellness program, accelerometer, incentives), where only intervention participants will receive reward points for completing daily step count goals.

After randomization, a baseline 'run-in' assessment phase will occur one week prior to the study intervention (T0). During this 'run-in' period, participants will wear a Bluetooth enabled StepsCount Piezo accelerometer, which will track participants' daily steps and moderate to vigorous physical activity (MVPA), and synchronize their accelerometer (i.e. upload information) to the Change4Life program for seven days. Participants will also be asked to complete the Behavioural Regulation to Exercise Questionnaire (BREQ-3) and the Self-Efficacy for Exercise Scale.

Throughout the 24-week study, all participants will be asked to wear the accelerometer and synchronize it to the Change4Life program daily. Date, steps per day, and bout minutes of MVPA per day (bouts include 10 or more continuous minutes of MVPA) will be collected when the accelerometer is synchronized. Daily synchronization from the accelerometer to the Change4Life program must be completed by 10 am the next morning. Participants will be instructed to increase their daily step counts by 1,000 and 2,000 steps above baseline (T0) over the course of the first six weeks of the study. On week 7, participants will be asked to increase daily steps per day to 3,000 over baseline, and maintain that level of activity for the duration of the study.

Outcome measures will be assessed at baseline (T0), intervention end point (T2), and follow up (T3).

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* English speaking

Exclusion Criteria:

* Existing medical condition, which could be exacerbated by physical activity as measured by the Physical Activity Readiness Questionnaire.

Note. Participants cannot enrol in the study without Internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Steps | Daily for 24 weeks
  Steps per day will be objectively assessed using the Bluetooth enabled, medical grade, StepsCount Piezo accelerometer

SECONDARY OUTCOMES:
10 Minute Bouts of Moderate to Vigorous Physical Activity | Daily for 24 weeks
  10 minutes bouts of moderate to vigorous physical activity per day will be objectively assessed using the Bluetooth enabled, medical grade, StepsCount Piezo accelerometer.
Motivation to Exercise - Behavioural Regulation to Exercise Questionnaire; BREQ-3 | Baseline (T0; week 0), intervention end point (T2; week 12), and follow up assessments (T3; week 24).
  Participants will be asked to complete the Behavioural Regulation to Exercise Questionnaire (BREQ-3; Markland & Tobin, 2004; Wilson et al., 2006), a 24-item questionnaire designed to measure self-determined motivation to exercise. This questionnaire will be administered online at baseline (T0; week 0), intervention end point (T2; week 12), and follow up assessments (T3; week 24).
Walking Self-Efficacy - Self-Efficacy for Exercise Scale; SEE Scale | Baseline (T0; week 0), intervention end point (T2; week 12), and follow up assessments (T3; week 24).
  Participants will be asked to complete a modified version of the Self-efficacy for Exercise (SEE) Scale (Resnick & Jenkins, 2000), a 9-item questionnaire designed to measure self-reported confidence to exercise (i.e. walk). This questionnaire will be administered online at baseline (T0; week 0), intervention end point (T2; week 12), and follow up assessments (T3; week 24).
10 Minute Bouts of Moderate to Vigorous Physical Activity | Intervention end point (T2; week 12), and follow up assessments (T3; week 24).
  Participants will also be asked to complete a modified version of the International Physical Activity Questionnaire - Short Form (IPAQ-SF), a six-item questionnaire designed to measure moderate and vigorous physical activity, as well as time spent walking (Booth, 2000; Craig et al., 2003). This questionnaire will be administered online at intervention end point (T2; week 12), and follow up assessments (T3; week 24).

CONTACTS AND LOCATIONS:
Overall Officials: Guy Faulkner, PhD, Principal Investigator — University of Toronto
Locations (1):
- Faculty of Kinesiology and Physical Education, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available

REFERENCES:
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] Markland D, Tobin V. A modification of the Behavioral Regulation in Exercise Questionnaire to include an assessment of amotivation. Journal of Sport and Exercise Psychology 26: 191-196, 2004.
- [Background] Wilson PM, Rodgers WM, Loitz CC, Scime G. "It's who I am…really!" The importance of integrated regulation in exercise contexts. Journal of Biobehavioral Research 11: 79-104, 2006.
- [Background] Booth M. Assessment of physical activity: an international perspective. Res Q Exerc Sport. 2000 Jun;71(2 Suppl):S114-20. No abstract available. PMID 10925833
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Derived] Mitchell M, White L, Oh P, Kwan M, Gove P, Leahey T, Faulkner G. Examining Incentives to Promote Physical Activity Maintenance Among Hospital Employees Not Achieving 10,000 Daily Steps: A Web-Based Randomized Controlled Trial Protocol. JMIR Res Protoc. 2016 Dec 12;5(4):e231. doi: 10.2196/resprot.6285. PMID 27956377